CLINICAL TRIAL: NCT05772923
Title: Organ Preservation in Patients With a Good Clinical Response After (Chemo)Radiation for Rectal Cancer: Defining the Role of Additional Contact X-ray Brachytherapy Versus Extending the Waiting Interval and Local Excision
Brief Title: Organ Preservation in Rectal Cancer: Contact X-ray Brachytherapy vs Extending the Waiting Interval and Local Excision
Acronym: OPAXX
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Netherlands Cancer Institute (Other)
Collaborators: Catharina Ziekenhuis Eindhoven (Other); ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M20PAX
Record Dates: First submitted 2021-03-04; First posted 2023-03-17 (Actual); Last update posted 2023-03-17 (Actual); Status verified 2023-03

CONDITIONS: Organ Preservation; Rectal Cancer; Quality of Life; Locally Advanced Rectal Carcinoma
Keywords: Organ preservation; Rectal cancer; (Chemo)radiation; Local excision; Contact x-ray brachytherapy; TAMIS
MeSH Terms: conditions — Rectal Neoplasms | interventions — Mastectomy, Segmental

STUDY DESIGN:
Intervention Model Description: This is a prospective study with a mixed design. It concerns a phase II feasibility study for patients in whom a good, but not complete response has been achieved after (chemo)radiation (OPAXX study): two parallel single study-arms evaluate the efficacy of experimental organ preservation approaches. To allow for a better comparison of secondary parameters (toxicity and morbidity of both additional local treatments) eligible patients will be randomized between two experimental arms. Furthermore, an observational cohort study is established to register rectal cancer patients with a good but not complete clinical response after (chemo)radiation who are not eligible for randomisation in the OPAXX study (OPAXX registration study).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Contact x-ray brachytherapy (Experimental): Contact x-ray brachytherapy will be given applied after randomisation with a maximum interval of 14 weeks after finishing the neoadjuvant (chemo)radiation. Contact x-ray brachytherapy consists of three fractions of 30Gy per fraction applied to the tumour, with a 2 week interval between each boost. Response evaluation takes place every 3 months thereafter. Patients in whom a clinical complete response is detected during follow-up are offered a watch-and-wait approach; patients in whom an incomplete response or disease progression is noted, completion or salvage TME-surgery is advised.
  Interventions: Radiation: Contact x-ray brachytherapy
- Extending the waiting interval, with or without local excision (Experimental): The waiting interval will be extended with 6-8 more weeks after the first response evaluation, followed by a second (or third in case of ongoing response) re-assessment. Patients with a clinical complete response at the time of the second (or third) response evaluation will be offered a watch-and-wait approach without any surgical treatment. Patients with a remaining small lesion will be offered transanal local excision. Depending on the final pathological staging after local excision, patients are categorized as low-risk or high-risk, and will be offered a watch-and-wait strategy or completion TME-surgery, respectively.
  Interventions: Procedure: Local excision

INTERVENTIONS:
Radiation: Contact x-ray brachytherapy — With contact x-ray brachytherapy an intraluminal radiation boost up to 90 Gy is applied to the primary rectal tumour, with minimal collateral damage to the surrounding normal tissues due to minimal penetration of the 50 kVolt therapy.
  Arms: Contact x-ray brachytherapy
Procedure: Local excision — Local excision will basically be performed by the TAMIS-procedure (transanal minimally invasive surgery).
  Arms: Extending the waiting interval, with or without local excision

SUMMARY:
The goal of this prospective phase II feasibility study is to evaluate two additional local treatment options in rectal cancer patients with a good clinical response after neoadjuvant (chemo)radiation: contact x-ray brachytherapy versus extension of the waiting interval with or without local excision, and to investigate which rate of organ preservation can be achieved.

DETAILED DESCRIPTION:
Rationale: The organ preservation approach for rectal cancer has been explored increasingly, aiming at improving quality of life by prevention of total mesorectal excision (TME-surgery). In patients with intermediate rectal cancer (IRC) and locally advanced rectal cancer (LARC) who receive neoadjuvant (chemo)radiotherapy (in general a short-course radiotherapy or a long-course chemoradiation, respectively) subsequent TME-surgery is still standard of care.

In patients with a good clinical response after neoadjuvant (chemo)radiation, organ preservation may be considered, depending on the extent of the response monitored by radiological and endoscopic assessment. Some patients show a clinical complete response and can be monitored closely in a watch-and-wait approach. In case of a good, but not complete response, it remains unclear which patients may benefit from extension of the observation period after (chemo)radiation in order to achieve a complete clinical response over time, or in whom additional local treatment options (such as contact x-ray brachytherapy or local excision) are beneficial in obtaining organ preservation eventually.

Objective: The aim of this study is to investigate which rate of organ preservation can be achieved in patients with rectal cancer treated with neoadjuvant (chemo)radiotherapy with a good clinical response, and to optimize the different treatment strategies. In patients with a near-complete response or a small residual tumour mass, participation is offered in a phase II feasibility trial, in which two potential organ preservation treatment strategies are evaluated: contact x-ray brachytherapy or extension of the waiting interval with or without additional local excision in case of residual disease.

Study design: This is a prospective study with a mixed design. It concerns a phase II feasibility study for patients in whom a good, but not complete response has been achieved after (chemo)radiation (OPAXX study): two parallel single study-arms evaluate the efficacy of experimental organ preservation approaches. To allow for a better comparison of secondary parameters (toxicity and morbidity of both additional local treatments) eligible patients will be randomized between two experimental arms. Furthermore, an observational cohort study is established to register rectal cancer patients with a good but not complete clinical response after (chemo)radiation who are not eligible for randomisation in the OPAXX study (OPAXX registration study).

Study population: In general, patients with IRC receiving short-course radiotherapy with delayed surgery (patients with initially a cT1-3, cN1-2 lymph nodal status, no involved MRF or cT3c-d, N0-1 lymph nodal status) or patients with LARC receiving neoadjuvant long-course chemoradiation (patients with initially cT4 tumour, cN2 lymph node status, lateral lymph node involvement and/or an involved mesorectal fascia (MRF+)) according to the Dutch national guideline are eligible for this study when at the first response assessment 6-8 weeks after finishing the (chemo)radiation a good clinical response is seen. A good clinical response has been defined as a clinical complete response, a near-complete response or a small residual tumour mass <3 cm on endoscopy, but also no evidence of residual nodal disease on magnetic resonance imaging (MRI) (ycN0). In case of a clinical complete response the current strategy of watchful waiting is offered. Eligible patients in whom a good, but not complete response is detected will be randomized to one of the two experimental OPAXX study arms, provided that both additional local treatment options are technically feasible.

Intervention arms OPAXX study:

Arm 1: Contact x-ray brachytherapy will be given applied after randomisation with a maximum interval of 14 weeks after finishing the neoadjuvant (chemo)radiation. Contact x-ray brachytherapy consists of three fractions of 30Gy per fraction applied to the tumour, with a 2 week interval between each boost. Response evaluation takes place every 3 months thereafter. Patients in whom a clinical complete response is detected during follow-up are offered a watch-and-wait approach; patients in whom an incomplete response or disease progression is noted, completion or salvage TME-surgery is advised.

Arm 2: The waiting interval will be extended with 6-8 more weeks after the first response evaluation, followed by a second (or third in case of ongoing response) re-assessment. Patients with a clinical complete response at the time of the second (or third) response evaluation will be offered a watch-and-wait approach without any surgical treatment. Patients with a remaining small lesion will be offered transanal local excision. Depending on the final pathological staging after local excision, patients are categorized as low-risk or high-risk, and will be offered a watch-and-wait strategy or completion TME-surgery, respectively.

Main study parameters/endpoints: The primary endpoint of the OPAXX study reflects the efficacy of both additional treatment options: the rate of successful organ preservation (defined as an in-situ rectum, no defunctioning stoma and absence of active locoregional cancer failure) at one year following randomisation in rectal cancer patients with a good, but not complete clinical response after (chemo)radiation. Secondary endpoints are related to toxicity and morbidity of the two additional treatment options in the randomisation study, as well as to oncological and functional outcomes at one, two and five years of follow-up.

For patients with a good but not complete clinical response after (chemo)radiation who are not eligible for randomisation in the OPAXX study an observational cohort study is conducted (OPAXX registration study).

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: Standard treatment of IRC and LAR consists of neoadjuvant short-course or long-course (chemo)radiotherapy followed by TME-surgery. If a clinical complete response is seen at response evaluation, a watch-and-wait approach is currently considered a valid strategy in selected patients according to the Dutch national guidelines. In the ongoing Dutch national prospective registry patients with a near-complete response are currently offered an extension of the observation period rather than TME-surgery, and, subsequently, a watch-and-wait policy when a clinical complete response is noted over time. On the other hand, all patients with a persistent residual lesion will proceed to TME-surgery.

In the current study, two experimental approaches are introduced that could increase organ preservation rates in patients with a good, but not-complete response at the first response evaluation: additional endoluminal contact x-ray brachytherapy and local excision of the tumour remnant.

Prior to randomisation, eligible patients are well informed about the risks of the two experimental treatment strategies (i.e. unclear long-term oncological outcome), and are offered standard-of-care TME-surgery. Moreover, patients will be informed that additional treatment with contact x-ray brachytherapy or local excision might increase the morbidity rates in case completion or salvage TME-surgery is required.

Finally, in both arms of this phase II study an intensive surveillance program has been established, in order to detect treatment failure, tumour regrowth or disease recurrence at an early stage, in order to proceed to completion or salvage TME-surgery when needed and when possible.

ELIGIBILITY:
Inclusion Criteria:

* histologically verified adenocarcinoma above the dentate line and within 10cm of the anal verge;
* neoadjuvant short-course radiotherapy for patients with 1) IRC and delayed response evaluation according to the Dutch national guidelines (cT1-3, cN1-2 lymph nodal status, no involved MRF or cT3c-d, N0-1 lymph nodal status without pres-ence of significant distant metastases) without full dose chemotherapy in the inter-val (e.g. Rapido-scheme) or 2) LARC due to comorbidity or frailty; OR
* neoadjuvant long-course radiotherapy (chemoradiation) for patients with 1) LARC according to the Dutch national guidelines (cT4 tumour, cN2 lymph nodal status, lateral lymph node involvement, and/or involved MRF, without the presence of significant distant metastases) or 2) early rectal cancer or IRC and a strong wish for organ preservation;
* clinically near-complete response or a small residual tumour mass <3 cm;
* technically feasible to perform both treatment options (contact x-ray brachytherapy or local excision);
* age >18 years;
* written informed consent.

Exclusion Criteria:

* neoadjuvant or induction chemotherapy prior or adjacent to (chemo)radiation, e.g. patients with a Rapido or M1-scheme are not eligible;
* radiation dose >50.4 Gy or boost dose on the primary tumour;
* presence of suspicious lymph nodes (yN1/N2) at first response evaluation;
* residual tumour ≥ 3cm or over half of the circumference of the rectal lumen;
* patients who are unable to undergo contact x-ray brachytherapy or local excision;
* patients who cannot tolerate a completion- or salvage-TME because of comorbidity or frailty;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Estimated)
Dates: Start 2021-04-16 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
Rate of successful organ preservation | At one year following randomisation
  Including an in-situ rectum (including patients subjected to local excision), no defunctioning stoma and absence of active loco-regional cancer failure (indicated as either local intraluminal tumour regrowth or regional recurrence in lymph nodes requiring TME-surgery)

SECONDARY OUTCOMES:
Incidence of radiation toxicity | Short-term (< 3 months after end of treatment) and long-term (< 12 months after end of treatment)
  Frequency of adverse events grade 3-4 defined by the common terminology criteria of adverse events (CTCAE) version 5.0
Incidence of postoperative morbidity after local excision | Short term (occurring within 3 months after local excision) and long-term (within one year)
  Frequency of post-operative complication grade 3-4 according to Clavien-Dindo
Frequency of patients with a high Low Anterior Rectal Syndrome (LARS) score | At baseline, at 3 months, one, two and five year
  Defined by the LARS questionnaire with a score between 30-42
Frequency of patients with impaired of bowel function | At baseline, at 3 months, one, two and five year
  Defined by an approved questionnaire IL108 from the European Organization for Research and Treatment of Cancer (EORTC) based on selected items of EORTC QLQ-PR25, QLQ-CX24 and QLQ-ANL27
Frequency of patients with impaired bladder function | At baseline, at 3 months, one, two and five year
  Defined by an approved questionnaire IL108 from the European Organization for Research and Treatment of Cancer (EORTC) based on selected items of EORTC QLQ-PR25, QLQ-CX24 and QLQ-ANL27
Frequency of patients with a minimum important difference (MID) of 5 to 10 points on health-related quality of life score (HRQoL-scores) | At baseline, at 3 months, one, two and five year
  Defined by the European Organization for Research and Treatment of Cancer (EORTC) QLQ-C29/30
Regrowth rate | At one- and two year
  Regrowth rate
Disease free survival | At one- and two year
  Disease free survival
Overall survival | At one- and two year
  Overall survival
Organ preservation rate | At two years
  Organ preservation rate
Number of patients with complications after completion or salvage TME-surgery | Within the first 30 days after surgery
  In terms of postoperative morbidity and mortality rates defined by Clavien-Dindo

CONTACTS AND LOCATIONS:
Overall Officials: Brechtje A Grotenhuis, MD, PhD, Principal Investigator — Antoni van Leeuwenhoek Hospital; Pim Burger, MD, PhD, Principal Investigator — Catharina Ziekenhuis Eindhoven
Locations (7):
- Netherlands (7):
  - Radbouw University Medical Centre, Nijmegen, Gelderland
  - Catharina Hospital, Eindhoven, North Brabant
  - Antoni van Leeuwenhoek, Amsterdam, North Holland
  - Deventer Hospital, Deventer, Overijssel
  - Isala, Zwolle, Overijssel
  - Medical Center Leeuwarden, Leeuwarden, Provincie Friesland
  - Ijsselland Hospital, Capelle aan den IJssel, South Holland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Geubels BM, van Triest B, Peters FP, Maas M, Beets GL, Marijnen CAM, Custers PA, Rutten HJT, Theuws JCM, Verrijssen AE, Cnossen JS, Burger JWA, Grotenhuis BA. Optimisation of Organ Preservation treatment strategies in patients with rectal cancer with a good clinical response after neoadjuvant (chemo)radiotherapy: Additional contact X-ray brachytherapy versus eXtending the observation period and local excision (OPAXX) - protocol for two multicentre, parallel, single-arm, phase II studies. BMJ Open. 2023 Dec 30;13(12):e076866. doi: 10.1136/bmjopen-2023-076866. PMID 38159950
- See also: study website — https://www.opaxx.nl/